CLINICAL TRIAL: NCT02685774
Title: A Randomized, Open-label, Single Dose, 2-way Crossover Study to Compare the Pharmacokinetic Characteristics of CKD-395 0.25/500 mg in Healthy Male Volunteers
Brief Title: A Clinical Study to Compare the Pharmacokinetic Characteristics of CKD-395 0.25/500mg in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 158BE15032
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT group (Other): R: Reference drug(Duvie Tab. 0.5mg 1T, Glucophage XR Tab. 500mg 2T) T: Test drug(CKD-395 0.25/500mg 2T)
  Interventions: Drug: Duvie Tab. 0.5mg, Glucophage XR Tab. 500mg; Drug: CKD-395 0.25/500mg
- TR group (Other): T: Test drug(CKD-395 0.25/500mg 2T) R: Reference drug(Duvie Tab. 0.5mg 1T, Glucophage XR Tab. 500mg 2T)
  Interventions: Drug: Duvie Tab. 0.5mg, Glucophage XR Tab. 500mg; Drug: CKD-395 0.25/500mg

INTERVENTIONS:
Drug: Duvie Tab. 0.5mg, Glucophage XR Tab. 500mg — Duvie Tab. 0.5mg 1T, Glucophage XR Tab. 500mg 2T oral administration
  Other Names: Duvie Tab. 0.5mg; Glucophage XR Tab. 500mg
Drug: CKD-395 0.25/500mg — CKD-395 0.25/500mg 2T oral administration

SUMMARY:
This study is a randomized, open-label, single dose, 2-way crossover study to compare the pharmacokinetic characteristics of CKD-395 0.25/500 mg in healthy male volunteers.

DETAILED DESCRIPTION:
To healthy male subjects of twenty six(26), following treatments are administered dosing in each period fed condition(high fat meals) and wash-out period is a minimum of 7 days.

Treatment A(Reference Drug): DuvieTM Tab. 0.5mg 1T + Glucophage XR Tab. 500mg 2T Treatment B(Test Drug): CKD-395 0.25/750mg Tab. 2T

Pharmacokinetic blood samples are collected up to 48hrs. Safety and pharmacokinetic are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy male whose age is over 19 years old when visiting for initial screening test
2. Body mass index (BMI) between 17.5 ~ 30.5 kg/m^2 and the body weight must be over 55kg

   * Body mass index (BMI) = weight (kg) / height (m)^2
3. A male with no congenital or chronic disease in three years, no history of symptoms in internal treatment, or no knowledge in the area
4. Due to the special characteristics of drugs, the participators must be qualified to do the clinical screening after examined through hematology test and blood chemistry analysis, urinary test, the electrocardiogram (ECG), and etc.
5. The participants must be volunteered and sign in an informed consent document proven by Chonbuk National University IRB before joining a study to show that he was given informed the purpose of tests and the special characteristics of drugs.
6. The participants must have an ability and willingness to participate throughout the entire trials

Exclusion Criteria:

1. A person who had a history or symptoms of clinically aware of blood, kidney, internal secretion, gastrointestinal, urinary system, cardiovascular, liver, mental, nervous, or allergic (except subclinical seasonal allergies that is not treated at injection) disease.
2. Who had a history of gastrointestinal related disease which can be affected the drug absorption (esophageal achalasia, esophagostenosis, esophageal disease, or Crohn's disease) or surgeries (except a simple appendectomy or herniotomy)
3. Who had following results after examination

   a. ALT or AST > twice higher than normal value
4. Who constantly intake 210 g/week of alcohol within 6 months of the screening. (a cup of beer (5%) (250mL) = 10 g, a shot of soju (20%) (50mL) = 8 g, a glass of wine (12%) (125 mL) = 12 g)
5. Who participated other clinical test or took testing bioequivalence drugs in 3 months before the first clinical drug trial
6. Whose blood pressure > 140 mmHg (systolic blood pressure) or > 90 mmHg (diastolic pressure)
7. Who had a medical history of alcohol and drug abuses.
8. Who had taken a drug that has a control of metabolic rate (activation or inhibition) in 30 days before the first taking of clinical testing drug
9. Who smokes more than 20 cigarettes per day
10. Who took prescribed drugs or over-the-counter drugs in 10 days before taking of very first clinical testing drug
11. Who participated in whole blood donation in 2 months before the first taking of clinical testing drugs or platelet donations in 1 month before the first taking to clinical testing drugs.
12. Who has a potent to increase a danger by participating in the clinical trials or who can interrupt interpreting test results by having serious or chronic medical and mental status or having issues in results of the screening examination.
13. Who has a history of an extreme sensitivity of drugs that contain Rosiglitazone or drugs that have similar effect as Rosiglitazone (Pioglitazone), or drugs that contain the ingredients of Metformin or biguanidine drugs
14. Who has a serious heart failure or a congestive heart failure that must be drug-treated
15. A patient with hepatopathy
16. A patient with severe nephropathy
17. Who has diabetic ketoacidosis or a diabetic coma, or type 1 diabetes, or has history of acute metabolic acidosis or ketoacidosis
18. A patient with serious infectious disease or severe injuries before and after a surgery
19. Who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders
20. A patient who has kidney disease or renal insufficient that are caused by cardiovascular collapse (shock) and acute myocardial infarction (a male with higher serum creatinine of 1.5mg / dL, or less creatinine clearance of 80 mL / min)
21. A patient who is being tested to inject radiological iodine contrast agent into blood vessels (ex: intravenous urography, intravenous cholangiography, angiography, using contrast medium computer tomography, etc.)
22. Who has severe systematic infection or severe trauma
23. Who has nutritional status, starvation, debilitating condition, pituitary dysfunction, or adrenal insufficiency patients
24. Who has respiratory dysfunction, gastrointestinal disease
25. Who is unable to take high fat foods
26. Who cannot limit intake of grapefruit or grapefruit containing foods in 7 days from the first dosing of clinical testing drug to collect pharmacokinetic blood samples
27. Test subjects who is not willing or unable to comply with guidelines described in this protocol
28. A person who is not determined unsuitable to participate in this test by the researchers

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
AUClast of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
Cmax of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
AUClast of Metformin | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs
Cmax of Metformin | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs

SECONDARY OUTCOMES:
AUCinf of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
Tmax of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
t1/2 of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
CL/F of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
Vd/F of Lobeglitazone | 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs
AUCinf of Metformin | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs
Tmax of Metformin | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs
t1/2 of Lobeglitazone | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs
CL/F of Metformin | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs
Vd/F of Metformin | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24 and 48hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No